CLINICAL TRIAL: NCT02177565
Title: Autologous Stem Cell Therapy for Fracture Non-union Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government)
Collaborators: Keele University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RL1 254; Issuing Organisation (Other: Robert Jones & Agnes Hunt Orthopaedic Hospital)
Record Dates: First submitted 2014-06-20; First posted 2014-06-27 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2014-06

CONDITIONS: Non-union of Fractures
Keywords: Non-union; fracture; bone marrow stem cells
MeSH Terms: conditions — Fractures, Bone | interventions — Carrier State

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- carrier plus BMSCs (Experimental): carrier plus in vitro expanded autologous BMSCs
  Interventions: Biological: carrier plus in vitro expanded autologous BMSCs
- carrier alone (control). (Placebo Comparator): Carrier alone
  Interventions: Biological: carrier plus in vitro expanded autologous BMSCs

INTERVENTIONS:
Biological: carrier plus in vitro expanded autologous BMSCs — The non-unions of fractures were stabilized with internal or external fixation devices. The non-union site was clearly exposed and decorticated to introduce sub-periosteal bone graft. Depending on the surgical approach, the site was partitioned in either medial/lateral or anterior/posterior sides. The contents of each universal container were mixed individually with a carrier by the surgeon, who was blinded to the contents of the container

SUMMARY:
Do mesenchymal stem cells accelerate new bone formation in persistent non-unions.

DETAILED DESCRIPTION:
Do mesenchymal stem cells accelerate new bone formation in persistent non-unions treated with carrier plus in vitro expanded autologous BMSCs or carrier alone (control). Secondary aims were to analyze predictors of union in these patients and describe adverse events at final follow-up.

ELIGIBILITY:
Inclusion Criteria:

* An established non-union according to the US Food & Drug Administration criteria14.
* Non-union following fracture of tibia or femur suitable for synthetic bone grafting.

Exclusion Criteria:

1. Skeletal immaturity.
2. Pregnant or breast-feeding.
3. Non-union following pathological fractures.
4. Positive to Hepatitis B, Hepatitis-C or HIV.
5. Infection during BMSC culture.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2000-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Radiological assessment of new callus and fracture bridging | 12 months
  The primary outcome measure was formation of new callus and cortical bridging, assessed from pre-operative and multiple post-operative radiographs and CT-scans up to 12 months. These images were divided into early (0-3 months) and late (9-12 months) groups. Non-unions were assessed from anonymized slides by four independent reviewers (two radiologists and two orthopedic surgeons) blinded to the side of cell insertion. Each slide had a pre-operative radiograph for comparison but no indication of time since surgery, and showed a medial/ lateral or an anterior/ posterior view depending on the surgical approach . At first, each reviewer indicated the side with largest callus and most cortical bridging pre-operatively. Then each reviewer examined subsequent radiographs to indicate the side with the largest increase in new callus and cortical bridging.

SECONDARY OUTCOMES:
EQ-5D | 12 months
  Change in EQ-5D index at 1 year was used as secondary outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: James Richardson, FRCS MD, Principal Investigator — Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust
Locations (1):
- Robert Jones & Agnes Hunt Orthopaedic Hospital, Oswestry, Shropshire, United Kingdom